CLINICAL TRIAL: NCT04760067
Title: Comparison of Sport Injury Anxiety of Athletes Doing Sports on Different Surfaces
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Other Study IDs: KaratayUH1
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-02

CONDITIONS: Athletic Injuries
Keywords: Sports injuries; Anxiety; Surface
MeSH Terms: conditions — Athletic Injuries; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Turf: After obtaining the demographic information of the athletes participating in our study, information about injury anxiety and injury anxiety will be collected with the Sports Injury Anxiety Scale.
  Interventions: Other: Sports Injury Anxiety Scale
- Artificial Turf: After obtaining the demographic information of the athletes participating in our study, information about injury anxiety and injury anxiety will be collected with the Sports Injury Anxiety Scale.
  Interventions: Other: Sports Injury Anxiety Scale
- Wood Parquet: After obtaining the demographic information of the athletes participating in our study, information about injury anxiety and injury anxiety will be collected with the Sports Injury Anxiety Scale.
  Interventions: Other: Sports Injury Anxiety Scale

INTERVENTIONS:
Other: Sports Injury Anxiety Scale — Sports Injury Anxiety Scale

SUMMARY:
Due to its nature, sports are an activity in which injuries are common. Sports injuries have athletic and environmental reasons. In sports injuries, although the medical team is generally interested in the physiological aspect of the injury, in recent years, the psychological aspect of the injury has also started to be taken care of. One of these psychological aspects is anxiety. Athletes who develop sports injury anxiety are more prone to injury. One of the environmental reasons is the ground for sports. We could not find a study in the literature comparing the anxiety levels of those who do sports on different grounds in different sports branches. Our study will provide support to the literature in this direction.

DETAILED DESCRIPTION:
The study will be carried out on volunteers after the approval of the ethics committee. Before the research, individuals and / or their relatives will be informed about the purpose and content of the study. Volunteer athletes between the ages of 18-35 without any known health problems will be included in the study after obtaining their informed consent.

150 athletes competing on turf, artificial turf and wooden parquet will be included in our study.

The data of our study will be collected by Google survey. After obtaining the demographic information of the athletes participating in our study, the data on injury anxiety will be collected with the Sports Injury Anxiety Scale.

ELIGIBILITY:
Inclusion Criteria:

* To be a healthy, previous injury athlete

Exclusion Criteria:

* Have an ongoing injury

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Healthy athletes with a history of injury
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-05-09 (Actual)

PRIMARY OUTCOMES:
Sports Injury Anxiety | Baseline
  It will be implemented to identify athletes' injury anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan GERÇEK, Principal Investigator — KTO Karatay Üniversitesi
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)